CLINICAL TRIAL: NCT04415177
Title: Safety and Effectiveness of Virtual Reality Utilizing EaseVRx for the Reduction of Chronic Pain and Opioid Use
Brief Title: Virtual Reality Trial Using EaseVRx For Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AppliedVR Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-521
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Chronic Lower Back Pain
Keywords: Virtual Reality; Chronic Lower Back Pain; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR Program A (Experimental): Software with active intervention
  Interventions: Device: EaseVRx headset with active intervention
- VR Program B (Active Comparator): Software without active intervention
  Interventions: Device: EaseVRx headset without active intervention

INTERVENTIONS:
Device: EaseVRx headset with active intervention — VR software developed by AppliedVR informed by evidence-based cognitive behavioral therapy principles, biofeedback and mindfulness strategies for pain management.
  Arms: VR Program A
Device: EaseVRx headset without active intervention — VR software developed by AppliedVR with neutral non-interactive content.
  Arms: VR Program B

SUMMARY:
Randomized, 2-arm parallel group clinical trial evaluating the effectiveness of a self-administered Virtual Reality program for the treatment of chronic lower back pain compared to a placebo VR program.

DETAILED DESCRIPTION:
A randomized, 2-arm parallel-group clinical trial evaluating the effectiveness of a self-administered Virtual Reality (VR) program for the treatment of chronic lower back pain. The primary objective of this study is to assess the impact of skills-based VR on changes in patient-reported pain and pain interference over the course of an 8-week intervention as well as compared to a placebo VR condition. The secondary objective is to assess the impact of skill-based VR on changes in patient-reported satisfaction over the course of an 8-week intervention and compared to a placebo VR condition. A tertiary objective is to assess the impact of skills-based VR on changes in patient-reported opioid use, physical function, behavioral skills development, and health outcomes immediately following the intervention relative to a pre-intervention baseline and compared to a placebo VR condition. An exploratory objective is to assess the impact of skills-based VR on changes in patient-reported pain levels, opioid use, physical function, behavioral skills development, health outcomes, and satisfaction at the 24-week post-intervention time point and compared to a placebo VR condition.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-85 years old
* Diagnosis of low back pain without radicular symptoms
* Pain duration of at least 6 months
* Average pain intensity of at least 4 on the 0-10 DoD/VA Pain Scale for the past month at screening
* English fluency
* Willing to comply with study procedures/restrictions

Exclusion Criteria:

* Unable to understand the goals of the study due to cognitive difficulty
* Current or prior diagnosis of epilepsy, seizure disorder, dementia, migraines or other neurological disease that may prevent the use of VR
* Medical condition predisposing to nausea or dizziness
* Hypersensitivity to flashing light or motion
* No stereoscopic vision or severe hearing impairment
* Injury to eyes, face or neck that prevents comfortable use of VR
* Pain related to cancer
* Active suicidal ideation or severe depression
* Previous use of EaseVR for pain
* Current participation in any interventional research study or completed participation in past 2 months
* Currently pregnant or planning to become pregnant
* Does not have access to WIFI during participation in study
* Currently works at or has an immediate family member who works for a digital health company or pharmaceutical company that provides treatments for acute or chronic pain

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Department of Defense (DoD)/VA Pain scale | The primary efficacy endpoint is the change from study baseline to Day 56
  DoD/VA Pain scale measures pain intensity, and inference around activity, sleep, mood, and stress, each on an 11-point scale. The max score is 50 and the minimum is 0. The higher the score the worse the outcome. This will be assessed twice weekly during the 8-week intervention intervention period.

SECONDARY OUTCOMES:
Patient's Global Impression of Change Scale | twice weekly during 8-week intervention, Day 56
  Single item Patient's Global Impression of Change Scale (PGIC), self-reported the level of change (if any) in activity limitations, symptoms, emotions, and overall quality of life-related to your painful condition on a 7-point scale. The higher the number the better the outcome.

OTHER OUTCOMES:
Device utilization Questionnaire | twice weekly during 8-week intervention, Day 56
  Self-reported number of VR sessions completed since the participant last reported. The scale is 0-4 or more. The higher than number the higher the usage.
VR Satisfaction Scale | Day 56
  Satisfaction ratings regarding the ability of the VR program to relieve pain symptoms on a 5-point scale. One is defined as strongly disagree with the statement and five is defined as strongly agree. The higher the number the better the outcome.
Custom Opioid Use Survey | Baseline, Day 56
  Custom survey assesses the use of opioids, frequency of use, dose of medication, happiness with regimen, and interest in change in treatment.
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function | Baseline, Day 56
  This 6-item PROMIS physical function measure assesses physical function such as (chores, running errands) on a 5-point scale. The max score is 30 and the minimum is 6. The higher the score the better the outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance | Baseline, Day 56
  6-item PROMIS sleep disturbance measure assesses the level of sleep disturbance on a 5-point scale. The max score is 30 and the minimum is 6. The higher the score the worse the outcome.
Pain Self-efficacy Questionnaire | Baseline, Day 56
  2-item PSEQ (PSEQ-2) assesses pain self-efficacy on a 7-point scale. The max score is 12 and the minimum is 0. The higher the score the better the outcome.
Pain Catastrophizing Scale | Baseline, Day 56
  4 items from the Pain Catastrophizing Scale (PCS) assesses frequency of pain-related thoughts and feelings on a 5-point scale. The max score is 16 and the minimum is 0. The higher the score the worse the outcome.
Chronic Pain Acceptance Questionnaire | Baseline, Day 56
  8-item Chronic Pain Acceptance (CPAQ-8) questionnaire assesses acceptance or psychological flexibility associated with chronic pain on a 7-point scale. The max score is 56 and the minimum is 8. The higher the score the better the outcome.
Behavioral Skills Assessment | Day 56
  Custom survey assesses the development of skills to manage pain outside of the VR headset. This is only included in the EaseVRx condition. There are 4 knowledge questions. These are on a 1-5 scale from do not agree to completely agree. The skills questions are on a 0 to 10 scale with 0 being not at all confident and 10 being very confident.
Health Utilization Outcomes Questionnaire | Day 56
  Questionnaire on the frequency of steroid injections, lower back surgery, emergency department visits, hospital admissions, and unplanned physician visits over various time periods. The first part of each of these questions asks if they have had the service and then the second part asks for the frequency.
VR Use Data | Day 1 through Day 56
  VR use calculated as the total number of sessions launched. It will be continuous data stored on the headset.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Garcia, PhD, Principal Investigator — AppliedVR Inc.
Locations (1):
- AppliedVR, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia L, Birckhead B, Krishnamurthy P, Mackey I, Sackman J, Salmasi V, Louis R, Castro C, Maddox R, Maddox T, Darnall BD. Durability of the Treatment Effects of an 8-Week Self-administered Home-Based Virtual Reality Program for Chronic Low Back Pain: 6-Month Follow-up Study of a Randomized Clinical Trial. J Med Internet Res. 2022 May 25;24(5):e37480. doi: 10.2196/37480. PMID 35612905
- [Derived] Garcia LM, Birckhead BJ, Krishnamurthy P, Mackey I, Sackman J, Salmasi V, Louis R, Maddox T, Darnall BD. Three-Month Follow-Up Results of a Double-Blind, Randomized Placebo-Controlled Trial of 8-Week Self-Administered At-Home Behavioral Skills-Based Virtual Reality (VR) for Chronic Low Back Pain. J Pain. 2022 May;23(5):822-840. doi: 10.1016/j.jpain.2021.12.002. Epub 2021 Dec 11. PMID 34902548
- [Derived] Garcia LM, Birckhead BJ, Krishnamurthy P, Sackman J, Mackey IG, Louis RG, Salmasi V, Maddox T, Darnall BD. An 8-Week Self-Administered At-Home Behavioral Skills-Based Virtual Reality Program for Chronic Low Back Pain: Double-Blind, Randomized, Placebo-Controlled Trial Conducted During COVID-19. J Med Internet Res. 2021 Feb 22;23(2):e26292. doi: 10.2196/26292. PMID 33484240
- [Derived] Garcia LM, Darnall BD, Krishnamurthy P, Mackey IG, Sackman J, Louis RG, Maddox T, Birckhead BJ. Self-Administered Behavioral Skills-Based At-Home Virtual Reality Therapy for Chronic Low Back Pain: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jan 19;10(1):e25291. doi: 10.2196/25291. PMID 33464215
- See also: webpage to assess if the study is right for you — https://appliedvr.io/study-enrollment/